CLINICAL TRIAL: NCT01596049
Title: The Efficacy of a Self-fixating Mesh in Unilateral Open Inguinal Hernia Repair, in Comparison to the Standard Treatment in the Literature
Brief Title: The Efficacy of a Self-fixating Mesh in Unilateral Open Inguinal Hernia Repair
Status: Terminated | Type: Observational
Why Stopped: recruitment was not going well.
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: hernia313-11-RMBCTIL
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Primary Inguinal Hernia; Unilateral Hernia; Open Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Self-fixating Mesh: patients attributed to that arm, undergoing surgery of open inguinal unilateral hernia repair, using Self-fixating Mesh which is acceptable in the literature.
  Interventions: Device: Self-fixating Mesh

INTERVENTIONS:
Device: Self-fixating Mesh — Using Self-fixating Mesh for Inguinal Hernia Repair

SUMMARY:
This study's objective is to assess the efficacy of a Self-fixating mesh in the surgical repair of unilateral inguinal hernia, which is becoming the new standard of care in open surgical repair of inguinal hernia.

The study design is interventional, enrolling 300 patients above 18 years of age, admitted for elective repair in the surgical department of Rambam Medical Health Care Campus, an academic medical center.

The study will assess several outcomes including post-surgical pain, recurrence, quality of life and post surgical complications (e.g. wound infection, the formation of hematoma or seroma, etc).

DETAILED DESCRIPTION:
This study's objective is to assess the efficacy of a Self-fixating mesh in the surgical repair of unilateral inguinal hernia, which is becoming the new standard of care in open surgical repair of inguinal hernia.

The study design is interventional, enrolling 300 patients above 18 years of age, admitted for elective repair in the surgical department of Rambam Medical Health Care Campus, an academic medical center.

The study will assess several outcomes including post-surgical pain, recurrence, quality of life and post surgical complications (e.g. wound infection, the formation of hematoma or seroma, etc).

The data will be compared to the literature and will be statistically analysed. The follow-up for each patient will be two years.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing primary unilateral open Inguinal Hernia Repair .
* patients undergoing elective surgery.
* above the age of 18 years old

Exclusion Criteria:

* patients having repeated Inguinal Hernia.
* patients having bilateral Hernia.
* patients undergoing laparoscopic surgery.
* patients undergoing non-elective surgery.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who are undergoing Inguinal Hernia Repair Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2012-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Percentage of post operative inguinal Hernia recurrence. | 2 weeks, 3,6,12,24 months post-operative
Post-operative patient quality of life will be assessed using a validated questionnaire. | 2 weeks, 3,6,12,24 months post-operative
Pain will be assessed by NRS (Numerical Rating Scale) | 2 weeks, 3,6,12,24 months post-operative
Post-operative complications will be assessed using a validated questionnaire. | 2 weeks, 3,6,12,24 months post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Adel Abu_Salih, M.D, Principal Investigator — Rambam health care campus, Haifa, Israel
Locations (1):
- Rambam health care campus, Haifa, Israel